CLINICAL TRIAL: NCT01060423
Title: A Randomized Phase II Trial of Irinotecan Drug-eluting Beads Administered by Hepatic Chemoembolization With Intravenous Cetuximab (DEBIRITUX) Versus Systemic Treatment With Intravenous Cetuximab and Irinotecan in Patients With Refractory Metastatic Colorectal Cancer and K-ras Wild-type Tumours
Brief Title: TACE With Irinotecan Drug-eluting Beads and Intravenous (IV) Cetuximab in Refractory Colorectal Cancer
Acronym: DEBIRITUX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor subject enrolment
Sponsor: Hans-Joachim Schmoll, MD (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor-Investigator, Hans-Joachim Schmoll, MD, MD, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2009-014728-44
Record Dates: First submitted 2010-01-27; First posted 2010-02-02 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal; liver metastasis; KRAS wildtype; chemoembolization; irinotecan eluting beads
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hepatic TACE with irinotecan eluting beads and iv cetuximab (Experimental): Irinotecan drug-eluting beads administered by hepatic chemoembolization with intravenous cetuximab (DEBIRITUX)
  Interventions: Drug: Cetuximab; Device: Irinotecan eluting BEADS
- iv cetuximab and irinotecan (Active Comparator): systemic treatment with intravenous cetuximab and irinotecan
  Interventions: Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: Cetuximab — Starting dose of 400mg/m2, followed by weekly 250mg/m2
  Other Names: Erbitux
Drug: Irinotecan — Irinotecan 180 mg/m² to be administered every two weeks
  Arms: iv cetuximab and irinotecan
Device: Irinotecan eluting BEADS — A minimum of two treatments per lobe (four bi-weekly sessions in the event of bilobar disease) at week 0 and 4 with up to 4ml (100-300µm DC Bead loaded with up to 200mg irinotecan) will be scheduled (i.e. for bilobar disease right lobe: week 0, left lobe: week 2, right lobe: week 4 and left lobe: week 6: following toxicity and extending interval if toxicity seen).
  Other Names: DC Bead
  Arms: hepatic TACE with irinotecan eluting beads and iv cetuximab

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Irinotecan Beads in combination with intravenous cetuximab versus intravenous irinotecan in combination with intravenous cetuximab in the treatment of patients with unresectable liver metastases from colorectal cancer.

Secondary objectives are safety and tolerability of hepatic chemoembolization and the question if the addition of aprepitant to standard antiemetic prophylaxis in patients treated by hepatic chemoembolization is safe and will reduce the rate of acute and delayed nausea and emesis.

DETAILED DESCRIPTION:
About half of patients with newly diagnosed colorectal cancer will develop metastatic disease and, however, in spite of the significant progress in the therapeutical strategies for metastatic disease, virtually all patients will eventually succumb to their illness. Based on prior clinical data there is a good rationale for the expectation that the combination of systemic chemotherapy and arterial chemoembolization with drug eluting beads may be effective in the setting of patients with unresectable or chemorefractory liver metastases. The aim of this study is therefore to assess whether the combination of Irinotecan eluting beads and intravenous cetuximab is safe and effective in the treatment of patients with unresectable liver metastases from refractory colorectal cancer and will result in a prolongation of disease control when compared to standard systemic treatment with intravenous irinotecan and intravenous cetuximab. In this patient group, intravenous irinotecan plus intravenous cetuximab may represent the "standard of care", with a previously described activity. The patient group is defined in terms of pretreatment, and the scientific question is whether the way of irinotecan administration by eluting beads in feasible and somehow beneficial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of stage IV (UICC) colorectal cancer with unresectable liver metastases (primary tumour may be present) and k-ras wild-type tumours
2. Patients had been treated and shown to be refractory to 5-FU (Capecitabine allowed)/oxaliplatin and/or 5-FU/irinotecan. Prior therapy with VEGF-inhibitors (e.g bevacizumab) is allowed
3. Patients with at least one measurable liver metastasis, with size > 1cm (RECIST criteria)
4. Patients with liver only or liver dominant disease (defined as ≥ 50 % tumour burden confined to the liver)
5. Patients with a portal vein not interfering with transarterial chemoembolization (e.g. no thrombosis) as judged by the investigator
6. ECOG Performance status ≤ 2
7. Life expectancy > 3 months
8. Age ≥ 18 years.
9. At least 4 weeks since last administration of last chemotherapy and/or radiotherapy (bone metastases may be allowed)
10. Patients who received VEGF-inhibition (e.g. with bevacizumab) in prior therapy are eligible if stopped since 4-6 weeks before randomization
11. Haematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 75 x109/L
12. INR < 1.5 (patients on therapeutic anticoagulants are not eligible)
13. Adequate liver function as measured by serum transaminases (AST & ALT) ≤ 3 x ULN and total bilirubin ≤ 1.5 x ULN
14. Adequate renal function: Serum creatinine ≤ 1.5 x ULN
15. Normal level of serum magnesium
16. Women of child bearing potential and fertile men are required to use effective contraception (negative serum βHCG for women of child-bearing age
17. Signed, written informed consent

Exclusion Criteria:

1. Presence of CNS metastases
2. Contraindications to irinotecan therapy (Chronic inflammatory bowel disease and/or bowel obstruction, history of severe hypersensitivity reactions to irinotecan hydrochloride trihydrate)
3. Active bacterial, viral or fungal infection within 72 hours of study entry
4. Women who are pregnant or breast feeding
5. Allergy to contrast media
6. Presence of another concurrent malignancy. Prior malignancy in the last 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
7. Any contraindication for hepatic embolisation procedures:

   * Large shunt as determined by the investigator (pretesting with lung perfusion scan not required)
   * Severe atheromatosis
   * Hepatofugal blood flow
8. Other significant medical or surgical condition, or any medication or treatment, that would place the patient at undue risk, that would preclude the safe use of chemoembolization or would interfere with study participation
9. Known hypersensitivity or contraindication to the drugs used in the trial (eg: cetuximab, 5-HT3 receptor antagonist, dexamethasone, or any component of aprepitant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate | 6 months after first administration of study medication

SECONDARY OUTCOMES:
Tumour Response (according to RECIST v1.1) | every three months up to progression of disease, maximum 12 months from the date of patient enrolment
  extent of treated lesions
Time to progression | every three months, until death of patient, maximum 12 months from the date of patient enrolment
Number of adverse events in study patients | whole study, every two weeks until 28 days from the date of last administration of study medication
Local tumour response | every three months up to progression of disease, maximum 12 months from the date of patient enrolment
  extent of necrosis in the treated lesions
Overall survival | every three months, until death of patient, maximum 12 months from the date of last patient enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Arnold, MD, Principal Investigator — Universitätsklinikum Eppendorf, Universitäres Cancer Center
Locations (13):
- Germany (13):
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Dresden
  - Zentralklinik Bad Berka GmbH, Abteilung für Interventionelle Radiologie, Bad Berka
  - Kliniken Essen-Mitte, Klinik für Innere Medizin IV, Essen
  - Klinikum Esslingen, Klinik für Onkologie, Gastroenterologie und Allgemeine Innere Medizin, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt/M.
  - Universitätsklinikum der Johann Wolfgang Goethe Universität Frankfurt, Frankfurt/M.
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - SLK-Kliniken Heilbronn, Heilbronn
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Medizinische Klinik und Poliklinik II, Tübingen
  - Universitätsklinikum Würzburg, Institut für Röntgendiagnostik, Würzburg